CLINICAL TRIAL: NCT01363843
Title: Complete Neoadjuvant Treatment for REctal Cancer (CONTRE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: William Sikov MD (Other)
Collaborators: Memorial Hospital of Rhode Island (Other); Rhode Island Hospital (Other); The Miriam Hospital (Other)
Responsible Party: Sponsor-Investigator, William Sikov MD, Prinicipal Investigator, Brown University
Organization: Brown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 224
Record Dates: First submitted 2011-05-26; First posted 2011-06-02 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: neoadjuvant; chemo/radiation; rectal cancer; rectum cancer; colon cancer; colorectal cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — Folfox protocol; Oxaliplatin; Leucovorin; Fluorouracil; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): Induction therapy - Modified FOLFOX6 - Oxaliplatin 85 mg/m2 + Leucovorin 400 mg/m2 IV, followed by 5-FU 400 mg/m2 IV, followed 5-FU 2400 mg/m2 IV by continuous infusion over 46 hours - Repeat q14 days x 8 cycles
  Concurrent Chemoradiation
  50.4 Gy Radiation in 28 fractions (45 Gy IMRT, 5.4 Gy 3D conformal boost)
  Surgery
  Interventions: Drug: FOLFOX6; Radiation: RT with concurrent chemotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: FOLFOX6 — FOLFOX6
  Other Names: Oxaliplatin 85 mg/m2; Leucovorin 400 mg/m2 IV; 5-FU 400 mg/m2 IV followed 5-FU 2400 mg/m2 IV by continuous over 46 hours
Radiation: RT with concurrent chemotherapy — IMRT 50.4Gy with chemotherapy
Procedure: Surgery

SUMMARY:
The purpose of this study is to find out how well patients with cancer of the rectum do if they get all of their other treatment - chemotherapy by itself followed by chemotherapy and radiation together - before surgery. Patients have recently been diagnosed with rectal cancer, and the doctors have recommended neo-adjuvant chemo treatment to try to shrink the cancer before removing it.

DETAILED DESCRIPTION:
The goals of treatment of locally advanced (T3-4 or N1-2) rectal cancer are to eliminate the primary tumor and any involved adjacent lymph nodes, minimize the risk of distant recurrence, and, when possible, preserve anal sphincter function. Standard treatment consists of surgery, concurrent chemotherapy and radiation (RT) and adjuvant chemotherapy. As the present time, the chemoradiation portion of the treatment is often administered before, as opposed to following, surgical resection. This approach has been associated with tumor down-staging, leading to higher rates of tumor resectability and an increase in the ability to perform sphincter-saving surgeries. (1). However, while advances in treatment of the primary tumor and regional nodes, specifically administration of preoperative chemoradiation and more aggressive surgical approaches, such as total mesorectal excision (TME), have been shown to improve locoregional disease control, toxicities and complications of these treatments may result in delay or omission of adjuvant chemotherapy, which could increase the risk of distant recurrence. In this pilot study, standard adjuvant chemotherapy (8 cycles of modified FOLFOX6) will be administered prior to chemoradiation and definitive surgery, eliminating the need for post-operative systemic therapy. The investigators will evaluate the ability of patients to tolerate this treatment and its impact on achievement of pathologic complete responses (pCRs), negative surgical margins and sphincter preservation.

ELIGIBILITY:
Inclusion Criteria

* Patients must have histologically proven adenocarcinoma of the rectum with no evidence of distant metastases.
* The tumor must be clinically Stage II (T3-4 N0 with N0 being defined as all imaged lymph nodes are < 1.0cm) or III (T1-4 N1-2 with the definition of a clinically positive node being any node > 1.0cm). Stage of the tumor may be determined by CT scan, endorectal ultrasound or MRI.
* Patients must have no evidence of distant metastases including liver metastases, peritoneal seeding, or inguinal lymphadenopathy.
* Patients must not have received prior chemotherapy or pelvic radiation for rectal cancer, or prior pelvic radiation for any other malignancy that would prevent the patient from receiving the required radiation treatments for this study.
* Patients must have a life expectancy of 5 years, excluding their diagnosis of cancer (as determined by the investigator).
* Patients must not have an active concurrent invasive malignancy. Patients with prior malignancies, including invasive colon cancer, are eligible if they are deemed by their physician to be at low risk for recurrence. Patients with squamous or basal cell carcinoma of the skin, melanoma in situ, carcinoma of the cervix, or carcinoma in situ of the colon or rectum that have been effectively treated are eligible, even if these conditions were diagnosed within 5 years prior to randomization.
* Patients must be > 18 years of age, ECOG performance status 0-1.
* ANC > 1,500/µl, platelets > 100,000/µl, total bilirubin < 2.0 mg/dl or direct bilirubin < 1.0 mg/dl, alkaline phosphatase < 3xULN, ALT < 3xULN, creatinine < 1.5xULN.
* The patient must have been evaluated by a surgeon, radiation oncologist and medical oncologist and all must concur that the patient is appropriate for this study.
* Signed informed consent; able to comply with study and/or follow- up procedures
* Peripheral neuropathy < grade 1

Exclusion Criteria:

* Evidence of metastatic disease.
* Rectal cancers other than adenocarcinoma, i.e., sarcoma, lymphoma, carcinoid, squamous cell carcinoma, cloacogenic carcinoma, etc.
* Pregnancy or lactation at the time of proposed randomization. Eligible patients of reproductive potential (both sexes) must agree to use adequate contraception.
* Any therapy for this cancer prior to randomization.
* Synchronous invasive colon cancer.
* Nonmalignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude the patient from receiving any chemotherapy treatment option or would prevent required follow-up.
* Patients with active inflammatory bowel disease, abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 6 months prior to Day 0 or other serious medical illness which might limit the ability of the patient to receive protocol therapy.
* Prior pelvic irradiation for any indication.
* Known hypersensitivity to 5-fluorouracil or oxaliplatin
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Sikov, MD, Principal Investigator — Brown University
Locations (3):
- United States (3):
  - Memorial Hospital, Pawtucket, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 39 patients we enrolled, 36 completed all 8 cycles of induction modified FOLFOX6, 35 patients completed chemo-radiation, 38 patients underwent surgery.
Groups:
- Study Arm Only: Induction therapy - Modified FOLFOX6 - Oxaliplatin 85 mg/m2 + Leucovorin 400 mg/m2 IV, followed by 5-FU 400 mg/m2 IV, followed 5-FU 2400 mg/m2 IV by continuous infusion over 46 hours - Repeat q14 days x 8 cycles
  Concurrent Chemoradiation with either continuous infusion 5-FU or capecitabine (MD choice)
  1. 5-FU 225 mg/m2 by continuous infusion starting the morning of the first dose of radiation and ending the morning after the last dose of radiation
  2. Capecitabine 825 mg/m2 PO BID
  50.4 Gy Radiation in 28 fractions (45 Gy IMRT, 5.4 Gy 3D conformal boost)
  Study Arm only (modified FOLFOX6): Induction;FOLFOX6 - Oxaliplatin 85 mg/m2 + Leucovorin 400 mg/m2 IV 5-FU 400 mg/m2 IV followed 5-FU 2400 mg/m2 IV by continuous over 46 hours q 14 days x 8 cycles Concurrent Chemoradiation with either continuous infusion 5-FU or capecitabine (MD choice)
  1. 5-FU 225 mg/m2 by continuous infusion(typical week of treatment is Monday AM thru Saturday AM = 1125 mg/m2/week)
  2. Capecitabine
Period: Overall Study
Arm/Group | Study Arm Only
Started | 39
Completed | 38 (39 enrolled, 36 completed 8 cycles of mFOLFOX6, 35 completed chemo-radiation, 38 underwent surgery.)
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Arm: Induction therapy - Modified FOLFOX6 - Oxaliplatin 85 mg/m2 + Leucovorin 400 mg/m2 IV, followed by 5-FU 400 mg/m2 IV, followed 5-FU 2400 mg/m2 IV by continuous infusion over 46 hours - Repeat q14 days x 8 cycles
  Concurrent Chemoradiation with either continuous infusion 5-FU or capecitabine (MD choice)
  1. 5-FU 225 mg/m2 by continuous infusion starting the morning of the first dose of radiation and ending the morning after the last dose of radiation
  2. Capecitabine 825 mg/m2 PO BID
  50.4 Gy Radiation in 28 fractions (45 Gy IMRT, 5.4 Gy 3D conformal boost)
  Study Arm only (modified FOLFOX6): Induction;FOLFOX6 - Oxaliplatin 85 mg/m2 + Leucovorin 400 mg/m2 IV 5-FU 400 mg/m2 IV followed 5-FU 2400 mg/m2 IV by continuous over 46 hours q 14 days x 8 cycles Concurrent Chemoradiation with either continuous infusion 5-FU or capecitabine (MD choice)
  1. 5-FU 225 mg/m2 by continuous infusion(typical week of treatment is Monday AM thru Saturday AM = 1125 mg/m2/week)
  2. Capecitabine
Arm/Group | Study Arm
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 61 [30 to 79]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Complete Resection
Description: The primary objective of this study is to determine the incidence of pCRs and complete (R0) resections at surgery after induction chemotherapy with 8 cycles of modified FOLFOX6 followed by standard chemoradiation with IMRT with concurrent infusional 5-FU or capecitabine
Time Frame: approx 6 months
Measure: Number; unit: participants
Arm/Group | Study Arm Only
Number analyzed (Participants) | 39
participants | 13

2. Secondary Outcome: Evaluate the Toxicity of Study Therapy
Description: Evaluate the toxicity of induction FOLFOX and subsequent infusional 5-FU or capecitabine/radiation. Results show number of patients who experienced a SAE. This does not mean all SAEs were deemed related to treatment.
  •Secondary efficacy measures include the clinical response rate, as measured endorectal ultrasound or pelvic MRI, and incidence and severity of toxicities seen during the various phases of study treatment, including treatment delays, bleeding and post-op complications. Each visit will have a toxicity assessment completed
Time Frame: approx 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Study Arm Only: Induction therapy - Modified FOLFOX6 - Repeat q14 days x 8 cycles
  Concurrent Chemoradiation with either continuous infusion 5-FU or capecitabine (MD choice)
  50.4 Gy Radiation in 28 fractions (45 Gy IMRT, 5.4 Gy 3D conformal boost)
  Study Arm only (modified FOLFOX6): Induction;FOLFOX6 - Oxaliplatin 85 mg/m2 + Leucovorin 400 mg/m2 IV 5-FU 400 mg/m2 IV followed 5-FU 2400 mg/m2 IV by continuous over 46 hours q 14 days x 8 cycles Concurrent Chemoradiation with either continuous infusion 5-FU or capecitabine (MD choice)
  1. 5-FU 225 mg/m2 by continuous infusion(typical week of treatment is Monday AM thru Saturday AM = 1125 mg/m2/week)
  2. Capecitabine
Arm/Group | Study Arm Only
Number analyzed (Participants) | 39
Participants | 13

ADVERSE EVENTS:
Time Frame: From signing consent to post completion of induction (approximately 4 months)
Description: induction AEs and SAEs included for reporting
Arm/Group | Study Arm Only
Serious Adverse Events (participants affected / at risk) | 13/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm Only (N=39)
anorexia (Investigations) | 1 (1)
angioderma/allergy (Investigations) | 1 (1)
constipation (Investigations) | 1 (1)
dehydration (Investigations) | 1 (1)
diarrhea (Investigations) | 2 (2)
DVT (Investigations) | 1 (1)
edema (Investigations) | 1 (1)
fever (Investigations) | 3 (3)
gastritis (Investigations) | 1 (1)
LFTs (Investigations) | 1 (1)
migrane/headache (Investigations) | 2 (2)
nausea (Investigations) | 3 (3)
neutropenia (Investigations) | 1 (1)
numbness (Investigations) | 1 (1)
pain-abdominal and cramps (Investigations) | 2 (2)
pain-neck (Investigations) | 1 (1)
Panic Attack (Investigations) | 1 (1)
parasthesia (Investigations) | 1 (1)
rash (Investigations) | 1 (1)
renal failure (Investigations) | 1 (1)
tingling (Investigations) | 1 (1)
thrombocytopenia (Investigations) | 1 (1)
thrombus formation (Investigations) | 1 (1)
TIA (Investigations) | 1 (1)
URI (Investigations) | 1 (1)
UTI (Investigations) | 1 (1)
vomiting (Investigations) | 2 (2)
weakness (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm Only (N=39)
Alk phos (Investigations) | 4 (4)
Albumin (Investigations) | 6 (6)
alopecia (Investigations) | 5 (5)
anemia (Investigations) | 21 (21)
anorexia (Investigations) | 6 (6)
anxiety (Investigations) | 4 (4)
vision disturbances (Investigations) | 4 (4)
pain-bone (Investigations) | 3 (3)
ca (Investigations) | 2 (2)
chills (Investigations) | 3 (3)
cold sensitivity (Investigations) | 11 (11)
constipation (Investigations) | 21 (21)
cough (Investigations) | 3 (3)
creatinine (Investigations) | 2 (2)
dehydration (Investigations) | 3 (3)
diarrhea (Investigations) | 16 (16)
dizziness (Investigations) | 6 (6)
dry skin, acne, itchiness, pruritus (Investigations) | 5 (5)
dyspnea/SOB (Investigations) | 5 (5)
dysuria (Investigations) | 2 (2)
edema (Investigations) | 3 (3)
fatigue (Investigations) | 31 (31)
heartburn (Investigations) | 2 (2)
bili (Investigations) | 2 (2)
glucose (Investigations) | 3 (3)
potassium (Investigations) | 9 (9)
Mg (Investigations) | 5 (5)
Hypersensitivity rxn (Investigations) | 4 (4)
hypertension/tach/palp (Investigations) | 5 (5)
HTN (Investigations) | 3 (3)
infection - general (tooth included here) (Investigations) | 2 (2)
insomnia (Investigations) | 4 (4)
LFTs (Investigations) | 10 (10)
light headedness (Investigations) | 2 (2)
mood alteration (Investigations) | 4 (4)
mucositis/oral thrush (Investigations) | 2 (2)
M/A (Investigations) | 2 (2)
nausea (Investigations) | 25 (25)
neuropathy (Investigations) | 19 (19)
neutropenia (Investigations) | 12 (12)
pain - mouth (Investigations) | 5 (5)
pain-abdominal and cramps (Investigations) | 7 (7)
pain-general (Investigations) | 3 (3)
pain-rectal (Investigations) | 7 (7)
palpatations/ tachycardia (Investigations) | 2 (2)
proteinuria (Investigations) | 2 (2)
rash (Investigations) | 5 (5)
rectal bleeding (Investigations) | 3 (3)
taste alteration (Investigations) | 5 (5)
thrombocytopenia (Investigations) | 18 (18)
uric acid (Investigations) | 2 (2)
urinary frequency (Investigations) | 3 (3)
vomiting (Investigations) | 8 (8)
WBC (Investigations) | 4 (4)
weight loss (Investigations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No